CLINICAL TRIAL: NCT05511402
Title: The Effect of Aerobic Training on Total Antioxidant Status, Total Oxidant Status, Glutathione, Oxidative Glutathione and Zonulin Levels in Patients With Parkinson's Disease
Brief Title: Effect of Aerobic Training on Oxidative Stress Markers in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Fatih Söke, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 630
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; exercise; total antioxidant status; total oxidant status; glutathione; oxidative glutathione; zonulin
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): This group will participate in an aerobic training program (8-week, 3 times weekly, and 30-min each time) and conventional physiotherapy program (8-week, 3 times weekly, and 45-min each time).
  Interventions: Other: Exercise training
- Conventional physiotherapy (Active Comparator): This group will participate in a conventional physiotherapy program (8-week, 3 times weekly, and 45-min each time).
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — People with Parkinson's Disease will be received a supervised physiotherapy and rehabilitation program.

SUMMARY:
Parkinson's disease is a chronic, neurodegenerative disorder characterized with the loss of dopamine-producing neurons. This loss is likely to be related with several environmental and genetic factors. One of the most important factor that is responsible for the initation and progression of the disease is oxidative stress. Exercise training, especially aerobic training, can change the levels of oxidative markers because exercise can lead to decrease oxidative stress in patients with Parkinson's disease. Therefore, this study aims to investigate (1) the effect of aerobic training on total antioxidant status, total oxidant status, glutathione, oxidative glutathione, and zonulin levels, (2) the relationship between the change of motor symptoms and disease severity and the change of total antioxidant status, total oxidant status, glutathione, oxidative glutathione, and zonulin levels.

ELIGIBILITY:
Inclusion Criteria:

* at least 40years of age
* diagnosed with Parkinson's Disease
* Hoehn and Yahr stage of 1 and 3

Exclusion Criteria:

* any other neurologic disorders,
* any cardiovascular, orthopedic, vestibular or rheumatic conditions that impact exercise training
* visual, auditory, and perception problems.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Total antioxidant status | 10 minutes
  Total antioxidant status is an important marker of total antioxidant capacity and it indicates an overall measure for the cumulative action of all antioxidants.
Total oxidant status | 10 minutes
  Total oxidant status is an significant marker of total oxidant capacity and it indicates an overall measure for the cumulative action of all oxidants.
Glutathione | 10 minutes
  Glutathione is an important intracellular antioxidant that protects against a variety of different antioxidant species.
Oxidative glutathione | 10 minutes
  Oxidative glutathione generated by glutathione reductase should be provided as decreased glutathione to the site.
Zonulin | 10 minutes
  The levels of zonulin can reflect systemic inflammation and oxidative stress.

SECONDARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale | 15 minutes
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale is the most commonly used scale to assess disease severity in Parkinson's Disease. It consists of four parts: (1) non-motor experiences of daily living, (2) motor experiences of daily living, (3) motor examination, and (4) motor complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Bora Tokcaer, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenner P. Oxidative stress in Parkinson's disease. Ann Neurol. 2003;53 Suppl 3:S26-36; discussion S36-8. doi: 10.1002/ana.10483. PMID 12666096
- [Background] Elokda A, DiFrancisco-Donoghue J, Lamberg EM, Werner WG. Effects of exercise induced oxidative stress on glutathione levels in Parkinson's disease on and off medication. J Neurol. 2010 Oct;257(10):1648-53. doi: 10.1007/s00415-010-5584-6. Epub 2010 May 12. PMID 20461398
- [Background] Dani C, Proenca IT, Marinho J, Peccin P, da Silva IRV, Nique S, Striebel V, Pochmann D, Elsner VR. Aquatic exercise program-modulated oxidative stress markers in patients with Parkinson's disease. Neural Regen Res. 2020 Nov;15(11):2067-2072. doi: 10.4103/1673-5374.276337. PMID 32394964
- [Background] Xu X, Fu Z, Le W. Exercise and Parkinson's disease. Int Rev Neurobiol. 2019;147:45-74. doi: 10.1016/bs.irn.2019.06.003. Epub 2019 Jun 20. PMID 31607362
- [Background] Khan Z, Ali SA. Oxidative stress-related biomarkers in Parkinson's disease: A systematic review and meta-analysis. Iran J Neurol. 2018 Jul 6;17(3):137-144. PMID 30886681
- [Background] Yuan Y, Tong Q, Zhang L, Jiang S, Zhou H, Zhang R, Zhang S, Xu Q, Li D, Zhou X, Ding J, Zhang K. Plasma antioxidant status and motor features in de novo Chinese Parkinson's disease patients. Int J Neurosci. 2016;126(7):641-6. doi: 10.3109/00207454.2015.1054031. Epub 2015 Jul 14. PMID 26010212
- [Background] Dumitrescu L, Marta D, Danau A, Lefter A, Tulba D, Cozma L, Manole E, Gherghiceanu M, Ceafalan LC, Popescu BO. Serum and Fecal Markers of Intestinal Inflammation and Intestinal Barrier Permeability Are Elevated in Parkinson's Disease. Front Neurosci. 2021 Jun 18;15:689723. doi: 10.3389/fnins.2021.689723. eCollection 2021. PMID 34220443
- [Background] Smeyne M, Smeyne RJ. Glutathione metabolism and Parkinson's disease. Free Radic Biol Med. 2013 Sep;62:13-25. doi: 10.1016/j.freeradbiomed.2013.05.001. Epub 2013 May 8. PMID 23665395
- [Background] Martin HL, Teismann P. Glutathione--a review on its role and significance in Parkinson's disease. FASEB J. 2009 Oct;23(10):3263-72. doi: 10.1096/fj.08-125443. Epub 2009 Jun 19. PMID 19542204